CLINICAL TRIAL: NCT00265915
Title: A CRC Trial of Rituximab in Combination With Sargramostim (GM-CSF) in Patients With Chronic Lymphocytic Leukemia
Brief Title: Rituximab and GM-CSF in Treating Patients With Chronic Lymphocytic Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: J0546 CDR0000450145; P01CA081534 (NIH); P30CA006973 (NIH); JHOC-J0546; JHOC-05070103; CLLRC-008
Record Dates: First submitted 2005-12-14; First posted 2005-12-15 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-08

CONDITIONS: Leukemia
Keywords: B-cell chronic lymphocytic leukemia; refractory chronic lymphocytic leukemia; stage 0 chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; sargramostim

INTERVENTIONS:
Biological: rituximab
Biological: sargramostim

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Colony-stimulating factors, such as GM-CSF, may increase the number of immune cells found in bone marrow or peripheral blood. Giving rituximab together with GM-CSF may be an effective treatment for chronic lymphocytic leukemia.

PURPOSE: This phase II trial is studying how well giving rituximab together with GM-CSF works in treating patients with B-cell chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the complete and overall response rate in patients with B-cell chronic lymphocytic leukemia treated with rituximab and sargramostim (GM-CSF).
* Determine the time to progression in patients treated with this regimen.
* Determine the effects of this regimen on CD20 antigen expression and soluble CD20 levels in these patients.

OUTLINE: This is a parallel-group, multicenter study. Patients are stratified according to disease status

Patients receive rituximab IV on days 4, 11, 18, and 25 and sargramostim (GM-CSF) subcutaneously on days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, 26, 29, 31, 33, 36, 38, 40, 43, 45, 47, 50, 52, and 54 (course 1). Patients with responding disease may receive an additional course of treatment.

After completion of study treatment, patients are followed periodically for up to 3 years.

PROJECTED ACCRUAL: A total of 130 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of B-cell chronic lymphocytic leukemia meeting 1 of the following criteria:

  * Previously treated stage III or IV or earlier stage disease with evidence of active disease, as defined by ≥ 1 of the following:

    * Weight loss > 10% within the past 6 months
    * Extreme fatigue
    * Fever or night sweats without evidence of infection
    * Worsening anemia or thrombocytopenia
    * Progressive lymphocytosis with a rapid lymphocyte doubling time
    * Marked hypogammaglobulinemia or paraproteinemia
    * Lymphadenopathy > 5 cm in diameter
  * Previously untreated stage 0-II disease with symptoms or significant fatigue or at high risk of progression due to of B2 microglobulin > 3.0 mg/mL
  * Patients who are ≥ 70 years of age with previously untreated stage III or IV or earlier stage disease requiring treatment but who refused chemotherapy are eligible

PATIENT CHARACTERISTICS:

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics

Hepatic

* Bilirubin < 2.0 mg/dL* (elevated bilirubin allowed if due to of Gilbert's disease) NOTE: *Liver dysfunction due to lymphocytic organ infiltration allowed

Renal

* Creatinine < 2.5 mg/dL* NOTE: *Renal dysfunction due to lymphocytic organ infiltration allowed

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active viral infection (e.g., viral hepatitis)

PRIOR CONCURRENT THERAPY:

Chemotherapy

* See Disease Characteristics

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2005-07; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Overall response rate

CONTACTS AND LOCATIONS:
Overall Officials: Ian W. Flinn, MD, PhD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins